CLINICAL TRIAL: NCT05608889
Title: Corrections Work's Adverse Effects and a Total Worker Health Program to Enhance Well-being
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kerry Kuehl (Other)
Responsible Party: Sponsor-Investigator, Kerry Kuehl, Professor of Medicine, Section Chief, and Director of Human Performance Laboratory, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-R2-CX-0006; 2020-R2-CX-0006 (Other Grant/Funding Number: U.S. Department of Justice (DOJ))
Record Dates: First submitted 2022-10-25; First posted 2022-11-08 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Occupational Stress; Health Behavior; Safety Issues; Mental Health Wellness 1
Keywords: Health Promotion; Mindfulness; Occupational Health; Total Worker Health; Safety
MeSH Terms: conditions — Occupational Stress; Health Behavior

STUDY DESIGN:
Intervention Model Description: This study will use a quasi-experimental pre-post design to compare values of outcome measures at the three times points: baseline, immediately post-intervention (3 months after baseline), and follow-up (9 months after baseline). Randomization of the intervention is not feasible at the individual level due to contamination effects within a site and no appropriate control condition. Furthermore, as each of the sites is unique, a randomized cluster design would not be able to account for confounders since there are only three sites, each with institutional differences. An advantage of the pre-post design is that each participant will act as their own control, increasing the power of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Enhanced Web App-enabled Total Worker Health Program (Experimental): The Total Worker Health Mindful Program will include 12, 45-minute sessions completed each week at participant's workplace. Sessions will be guided by written curriculum and focus on healthy eating, exercise, sleep and stress reducing behaviors enhanced by mindfulness activities. Participants will be provided with free enrollment codes to use the Headspace® application (app).
  Interventions: Behavioral: Total Worker Health Mindfulness Enhanced Program

INTERVENTIONS:
Behavioral: Total Worker Health Mindfulness Enhanced Program — The intervention will be delivered during 12, 45-minute weekly meetings of Correctional Professionals while on shift. Those sessions will be a combination of a video, mindfulness activity, and a group learning activity. It will conclude with members stating personal goals that will be followed up at the next meeting.
  Sessions will be scripted to make them easy to implement with high fidelity, and include tasks, learning activities, and wrap-up with practice instructions for each week. Coworkers will be responsible for running the sessions, which promotes shared norms and social support.

SUMMARY:
Conduct a quasi-experimental pre-post study of a mindfulness-enhanced, web/app-enabled, scalable Total Worker Health (TWH) program among higher stress Corrections Professionals. The primary outcomes relate to behaviors promoted by the program: being mindful/reduced stress/improved mood; healthier eating; more physical activity; greater restorative sleep; improved work-life balance and greater positive feelings about the organization.

DETAILED DESCRIPTION:
This proposed project will assess an innovative, scalable total worker health and wellness intervention among high stress Corrections Professionals. As stated in the proposal request, organizational and interpersonal factors have been associated with significant stress among Corrections Professionals, but there is limited assessment of effective and feasible interventions to mitigate these stress factors. Our current research has established robust constructs for characteristics of the organization and work environment, noting significant relationships with perceived stress. This critical understanding along with corresponding adverse mental and physical effects informs our proposed intervention to reduce potential stressors, enhance wellbeing, improve work performance, and reduce health care costs. This project will include a prospective interrupted time-series effectiveness trial of a mindfulness-enhanced, website/application-based, scalable Total Worker Health (TWH) program among higher risk corrections personnel working in restrictive housing units. Quantitative outcomes will include process measures; validated self-report indices of primary and secondary outcomes, and proximal potentially mediating factors; anthropometrics; laboratory studies of inflammation, vascular reactivity, and cellular aging; measures of job performance and health care costs. Qualitative measures will provide a deeper understanding of the quantitative findings. At program conclusion, there will be a cost effective easy to use work based health and wellness program tailored to corrections departments ready for dissemination. The robust dissemination plan includes coordinating the website and digital materials with the American Correctional Association marketing and media campaign site along with presentations at national corrections conferences making this freely available to all law enforcement and corrections personnel and agencies.

ELIGIBILITY:
Inclusion Criteria:

- Currently employed as a corrections professional at participating Oregon Department of Corrections facilities (Coffee Creek Correctional Facility and Oregon State Correctional Institution) for at least one month

Exclusion Criteria:

- Those who are not employed with participating Oregon Department of Corrections facilities listed above.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived stress | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Perceived Stress Scale Short Form (PSS-4)
Change in Mood | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  The Positive and Negative Affect Schedule (PANAS); Profile of Mood States Short Form (POMS-SF)
Change in Eating Habits | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Relevant excerpts from the National Cancer Institute's fruit and vegetable all day screener and Diet History Questionnaire (DHQ), percent calories from fat, and health dietary behaviors (Elliot et al., 2007; Kuehl et al., 2014)
Change in Physical Activity | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Change in physical activity will be assessed using this survey question: "How many days per week did you exercise or take part in moderate physical activities that increased your breathing a bit for a total of at least 30 minutes during the day (such as brisk walking or bicycling)?". This is measured in days per week (with a scale of 0-7 days). Relevant excerpts from previous research on physical activity behaviors (Elliot et al., 2007).
Change in Sleep | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Change in sleep will be assessed using this survey question: "In the past seven days, I had trouble sleeping" measures in a scale of 1-5 (1=very good, 2=good, 3=fair, 4=poor, 5=very poor). Short Form from the National Institutes of Health's Patient-Reported Outcomes Information System's Sleep Disturbance (PROMIS-SD-SF); Pittsburgh Sleep Quality Index (PSQI)
Change in Work-life balance | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Change in work-life balance will be assessed using this survey question: "In the past month, how often have you felt that you were able to control the important things in your life?" measured in a scale of 1-5 (1=none of the time, 2=a little of the time, 3=some of the time, 4=most of the time, 5=all of the time). Ballin et al., 2021.
Change in Feelings about organization | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Change in feelings about organization will be assessed using this survey question: "The Department of Corrections has processes in place that improve my work environment" measured with a scale from 1-5 (1=strongly disagree, 2=disagree, 3=neither disagree or agree, 4=agree, 5=strongly agree). Ballin et al., 2021.

SECONDARY OUTCOMES:
Change in Life Satisfaction | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Change in life satisfaction will be assessed with the survey question: "Would you say your general health is:" with a scale of a)excellent, b)very good, c)good, d)fair, and e)poor.
Change in Body Mass Index | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Change in Body mass index will measured in kg/m2.
Change in Blood Pressure | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Changes in blood pressure will be measured in mmHg.
Change in Vascular Reactivity | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Changes in Vascular reactivity will be measured in adjusted temperature rebound (aTR) between 0-2.
Change in C-reactive Protein | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Changes in C-reactive protein will be measured in mg/L.
Change in Cytokine Interleukin IL-6 | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Changes in cytokine Interleukin IL-6 will be measured in pg/mL.
Change in Tumour Necrosis Factor alpha | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Changes in Tumour Necrosis Factor alpha will be measured in pg/mL.
Change in telomere length | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Changes in telomere length will be measured in kb.
Change in Worker's Compensation Claims | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Change in Worker's Compensation Claims from Oregon Department of Corrections Human Resources data that report the number of worker's compensation claims there are.
Change in Days Injured | Change between timepoints: Before intervention implementation, 3 months after the intervention completion, and 9 months after intervention completion
  Change in Worker's Compensation Claims from Oregon Department of Corrections Human Resources data that report the number of missed days due to work-related illness or injury

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S. Kuehl, MD, DrPH, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon State Correctional Institute, Salem, Oregon
  - Coffee Creek Correctional Facility, Wilsonville, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliot DL, Goldberg L, Kuehl KS, Moe EL, Breger RK, Pickering MA. The PHLAME (Promoting Healthy Lifestyles: Alternative Models' Effects) firefighter study: outcomes of two models of behavior change. J Occup Environ Med. 2007 Feb;49(2):204-13. doi: 10.1097/JOM.0b013e3180329a8d. PMID 17293760
- [Background] Kuehl KS, Elliot DL, Goldberg L, MacKinnon DP, Vila BJ, Smith J, Miocevic M, O'Rourke HP, Valente MJ, DeFrancesco C, Sleigh A, McGinnis W. The safety and health improvement: enhancing law enforcement departments study: feasibility and findings. Front Public Health. 2014 May 8;2:38. doi: 10.3389/fpubh.2014.00038. eCollection 2014. PMID 24847475
- [Background] Cherniack M, Dussetschleger J, Dugan A, Farr D, Namazi S, El Ghaziri M, Henning R. Participatory action research in corrections: The HITEC 2 program. Appl Ergon. 2016 Mar;53 Pt A(Pt A):169-80. doi: 10.1016/j.apergo.2015.09.011. Epub 2015 Nov 2. PMID 26542616
- [Background] Creswell JD. Mindfulness Interventions. Annu Rev Psychol. 2017 Jan 3;68:491-516. doi: 10.1146/annurev-psych-042716-051139. Epub 2016 Sep 28. PMID 27687118
- [Background] Elliot DL, Mackinnon DP, Mabry L, Kisbu-Sakarya Y, Defrancesco CA, Coxe SJ, Kuehl KS, Moe EL, Goldberg L, Favorite KC. Worksite wellness program implementation: a model of translational effectiveness. Transl Behav Med. 2012 Jun;2(2):228-35. doi: 10.1007/s13142-012-0121-z. PMID 24073114
- [Background] Hammer LB, Ernst Kossek E, Bodner T, Crain T. Measurement development and validation of the Family Supportive Supervisor Behavior Short-Form (FSSB-SF). J Occup Health Psychol. 2013 Jul;18(3):285-96. doi: 10.1037/a0032612. Epub 2013 Jun 3. PMID 23730803
- [Background] Hammer LB, Truxillo DM, Bodner T, Rineer J, Pytlovany AC, Richman A. Effects of a Workplace Intervention Targeting Psychosocial Risk Factors on Safety and Health Outcomes. Biomed Res Int. 2015;2015:836967. doi: 10.1155/2015/836967. Epub 2015 Oct 18. PMID 26557703
- [Background] MacKinnon DP, Elliot DL, Thoemmes F, Kuehl KS, Moe EL, Goldberg L, Burrell GL, Ranby KW. Long-term effects of a worksite health promotion program for firefighters. Am J Health Behav. 2010 Nov-Dec;34(6):695-706. doi: 10.5993/ajhb.34.6.6. PMID 20604695
- [Background] Olson R, Wipfli B, Thompson SV, Elliot DL, Anger WK, Bodner T, Hammer LB, Perrin NA. Weight Control Intervention for Truck Drivers: The SHIFT Randomized Controlled Trial, United States. Am J Public Health. 2016 Sep;106(9):1698-706. doi: 10.2105/AJPH.2016.303262. Epub 2016 Jul 27. PMID 27463067
- [Background] Rohlman DS, Parish M, Elliot DL, Hanson G, Perrin N. Addressing Younger Workers' Needs: The Promoting U through Safety and Health (PUSH) Trial Outcomes. Healthcare (Basel). 2016 Aug 10;4(3):55. doi: 10.3390/healthcare4030055. PMID 27517968
- [Background] Tang YY, Yang L, Leve LD, Harold GT. Improving Executive Function and its Neurobiological Mechanisms through a Mindfulness-Based Intervention: Advances within the Field of Developmental Neuroscience. Child Dev Perspect. 2012 Dec;6(4):361-366. doi: 10.1111/j.1750-8606.2012.00250.x. PMID 25419230
- [Background] Uegaki K, de Bruijne MC, van der Beek AJ, van Mechelen W, van Tulder MW. Economic evaluations of occupational health interventions from a company's perspective: a systematic review of methods to estimate the cost of health-related productivity loss. J Occup Rehabil. 2011 Mar;21(1):90-9. doi: 10.1007/s10926-010-9258-0. PMID 20668923
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131
- [Background] Zweber ZM, Henning RA, Magley VJ. A practical scale for Multi-Faceted Organizational Health Climate Assessment. J Occup Health Psychol. 2016 Apr;21(2):250-9. doi: 10.1037/a0039895. Epub 2015 Nov 16. PMID 26569133
- [Derived] Elliot D, Kuehl K, DeFrancesco C, McGinnis W, Ek S, Van Horne A, Kempany KG. Technology-Enabled Intervention to Enhance Mindfulness, Safety, and Health Promotion Among Corrections Professionals: Protocol for a Prospective Quasi-Experimental Trial. JMIR Res Protoc. 2023 Sep 22;12:e45535. doi: 10.2196/45535. PMID 36602914
- See also: Ballin, J. , Niederhausen, M. , Kuehl, K. , Elliot, D. , McGinnis, W. and DeFrancesco, C. (2021) Defining Stress among Corrections Professionals. Open Journal of Preventive Medicine, 11, 237-250. doi: 10.4236/ojpm.2021.116019. — https://www.scirp.org/journal/paperinformation.aspx?paperid=109823